CLINICAL TRIAL: NCT04092413
Title: Subclinical Nail Involvement in Relevant Skin Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, YSAbdelraheem, principal investigator, Assiut University
Other Study IDs: SNIRSD
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Nail Diseases
MeSH Terms: conditions — Nail Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dermoscope — It is a non invasive tool that permits the visualization of morphological features that are not visible to the naked eye thus representing a link between macroscopic dermatopathology .

SUMMARY:
Onychopathies constitute one of the major challenges faced by a dermatologist in terms of its early detection and diagnosis .

Many disorders can affect the nails, including deformity and dystrophy, infections, and ingrown toenails. Infections can involve any part of the nail and may or may not change the nail's appearance. Most nail infections are fungal (onychomycosis), but bacterial and viral infections occur .

DETAILED DESCRIPTION:
Nails are characteristically affected in skin diseases such as psoriasis (speckling, psoriatic oil spot, crumbling nails, pachyonychia) ,lichen( anonychia, dystrophy) ,alopecia areata (speckling, trachyonychia, longitudinal grooves, leukonychia), atopic dermatitis (shiny nails, transverse grooves, speckling, paronychia) and other diseases.

Nail disorders are assessed by clinical inspection, dermatoscopy , microbiological (including mycological) testing, and histopathological examination by nail biopsy .

Utility of dermoscope as a tool for detection is increasing by the day and its use in onychopathies needs to be explored .

Nail dermoscopy has initially been used for the assessment of nail pigmentation . But its utilization has expanded for the diagnosis of all nail disorders; it became a routine diagnostic instrument, as its reveals helpful information. Dermoscopy can be applied to all visible parts of the nail unit, and even the nail matrix can be studied, in conjunction with intraoperative methods .

Nail dermoscopy offers many advantages. Mostly, it enhances visible nail features; however, it can also help identify additional unique and fascinating features, not visible to the naked eye. It is practical, noninvasive and still opens up a second microscopic level of inspection. It contributes toward confirmation of diagnosis and assessment of treatment response as well as prognosis.

In a cross-sectional study to detect signs of subclinical nail involvement in 68 patients with chronic plaque psoriasis, Forty-six patients showed nail dermoscopic findings. Coarse pits, onycholysis, oil drop sign and splinter hemorrhages were seen .

To the best of the investigator's knowledge, no available studies in the literature evaluate subclinical nail affection in skin diseases as lichen planus, atopic dermatitis and auto immune bullous diseases. Hence, with the help of a dermoscope,early diagnosis and appropriate treatment can be instituted.

ELIGIBILITY:
Inclusion Criteria:

- Patients complaining of common skin diseases ( psoriasis, atopic dermatitis, alopecia, lichen planus, and bullous diseases)

Exclusion Criteria:

* Patients who had gross visible nail changes will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients attending the Dermatology clinic , Assiut University Hospitals, Assiut, Egypt, during a period of one year complaining of ( psoriasis,PRP, lichen planus, atopic dermatitis and auto immune bullous diseases) will be recruited in the study
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subclinical nail involvement in relevant skin diseases | almost 6 months after start of the research
  dermoscopic examination of the nails searching for subclinical nail manifestations of some skin diseases like psoriasis , atopy , lichen , bullous diseases and alopecia areata

REFERENCES:
- [Background] Yadav TA, Khopkar US. Dermoscopy to Detect Signs of Subclinical Nail Involvement in Chronic Plaque Psoriasis: A Study of 68 Patients. Indian J Dermatol. 2015 May-Jun;60(3):272-5. doi: 10.4103/0019-5154.156377. PMID 26120154
- [Background] Tunc SE, Ertam I, Pirildar T, Turk T, Ozturk M, Doganavsargil E. Nail changes in connective tissue diseases: do nail changes provide clues for the diagnosis? J Eur Acad Dermatol Venereol. 2007 Apr;21(4):497-503. doi: 10.1111/j.1468-3083.2006.02012.x. PMID 17373977
- [Background] Nakamura RC, Costa MC. Dermatoscopic findings in the most frequent onychopathies: descriptive analysis of 500 cases. Int J Dermatol. 2012 Apr;51(4):483-5. doi: 10.1111/j.1365-4632.2010.04720.x. No abstract available. PMID 22435443
- [Background] Lencastre A, Lamas A, Sa D, Tosti A. Onychoscopy. Clin Dermatol. 2013 Sep-Oct;31(5):587-93. doi: 10.1016/j.clindermatol.2013.06.016. PMID 24079588
- [Background] Ronger S, Touzet S, Ligeron C, Balme B, Viallard AM, Barrut D, Colin C, Thomas L. Dermoscopic examination of nail pigmentation. Arch Dermatol. 2002 Oct;138(10):1327-33. doi: 10.1001/archderm.138.10.1327. PMID 12374538
- [Background] Grover C, Jakhar D. Onychoscopy: A practical guide. Indian J Dermatol Venereol Leprol. 2017 Sep-Oct;83(5):536-549. doi: 10.4103/ijdvl.IJDVL_242_16. PMID 28485306
- [Background] Jiaravuthisan MM, Sasseville D, Vender RB, Murphy F, Muhn CY. Psoriasis of the nail: anatomy, pathology, clinical presentation, and a review of the literature on therapy. J Am Acad Dermatol. 2007 Jul;57(1):1-27. doi: 10.1016/j.jaad.2005.07.073. PMID 17572277